CLINICAL TRIAL: NCT02163603
Title: A Multi-center Study on the Opportunity and Treatment of Residual Deformity After Reduction in Developmental Dislocation of the Hip
Brief Title: A Trial on the Opportunity and Treatment of Residual Deformity After Reduction in Developmental Dislocation of the Hip
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hongwen Xu (Other)
Collaborators: Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Hunan Children's Hospital (Other Government); Shenzhen Children's Hospital (Other Government); Foshan Hospital of Traditional Chinese Medicine (Other); Wuhan Women and Children's Medical Center (Other)
Responsible Party: Sponsor-Investigator, Hongwen Xu, Guangzhou Women and Children's Medical Center, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Other Study IDs: GuangzhouWCMC
Record Dates: First submitted 2014-05-06; First posted 2014-06-13 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Developmental Dislocation of the Hip; Congenital Dislocation of Hip; Residual Deformity; Reduction
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pelvic osteotomy
  Interventions: Procedure: Pelvic osteotomy

INTERVENTIONS:
Procedure: Pelvic osteotomy

SUMMARY:
Developmental dislocation of the hip is a common disease in children, and its incidence in China is about 9 ‰.The pathological changes of it is complex. The reluxation , subluxation and residual deformity and other complications are relatively common after treatment. The X-ray appears great acetabular index and wide medial gap , small central-edge angle. As there is no effective methods for treating such complications , investigators conducted this trial to find and prove optimal intervention time and treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria consists of patients with large acetabular index ,small central-edge angle after reduction in developmental dislocation of the hip

Exclusion Criteria:

* Age >14 years
* Patients are complicated with mental, neurological disorders (such as hypoxic-ischemic encephalopathy, epilepsy and dementia) or significant barriers to growth.
* Patients are complicated with cerebral palsy, multiple joint contractures disease.
* Children are complicated with dysfunction of liver and kidney , blood disorders, immune deficiency disease and ECG abnormalities.
* Parents refused further treatment.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The south of China
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Early treatment can achieve good results in the residual deformity after reduction in developmental dislocation of the hip | 3 years
  Acetabular index of all ages were measured ，and the acetabular index of patients getting early treatment (pelvis osteotomy ) is normal in all ages according to "The measurements of normal acetabular index and Sharp acetabular angle in Chinese hips" publised on Chinese Journal of Orthopaedics in 2010.